CLINICAL TRIAL: NCT01503671
Title: Effects of Atorvastatin Treatment on Left Ventricular Diastolic Function in Peritoneal Dialysis Patients (ALEVENT)
Brief Title: Effects of Atorvastatin Treatment on Left Ventricular Diastolic Function in Peritoneal Dialysis Patients
Acronym: ALEVENT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201108035MD
Record Dates: First submitted 2012-01-02; First posted 2012-01-04 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Heart Failure
Keywords: left ventricular diastolic function; inflammation; peritoneal dialysis; LV diastolic function changes after statin intervention
MeSH Terms: conditions — Heart Failure; Inflammation | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Experimental): Atorvastatin 40 mg/day for high inflammation CAPD patient
  Interventions: Drug: Atorvastatin
- No intervention arm (No Intervention): Placebo arm without intervention

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 40 mg/day
  Other Names: Lipitor
  Arms: Atorvastatin

SUMMARY:
Background

Heart failure is the final consequence of various heart disease and is also the leading cause of mortality worldwide. Diastolic dysfunction refers to an abnormality of diastolic distensibility, filling, or relaxation of the left ventricle. Patients with hypertensive left ventricular hypertrophy and an echocardiogram showing a normal ejection fraction and abnormal left ventricular filling can be said to have diastolic dysfunction. If pulmonary edema or effort dyspnea developed in such a patient. The term diastolic heart failure would be appropriate.

Pathology leading to diastolic heart failure include: impaired relaxation, increased passive stiffness, endocardial and pericardial disorders, microvascular flow and neurohormonal regulation. Among them, the association of pro-inflammatory system and diastolic dysfunction are already established. The investigators therefore hypothesized that the change of serum inflammatory markers might be associated with the change of left ventricular diastolic function and the investigators thus conducted a randomized case-control trial with this regard.

Method and materials

This is a case-control randomized study. The definition of left ventricular diastolic function is according to Guideline from the ACC and AHA. The investigators will evaluate left ventricular diastolic function noninvasively by echocardiography before and after the intervention. Exclusion criteria include coronary artery disease, significant valvular heart disease, cardiomyopathy, pericardial disease and renal insufficiency. The investigators would like to enroll 50 cases and the same numbers of the controls. The inclusion criteria are subjects who underwent peritoneal dialysis at the investigators hospital for more than 6 months with higher pro-inflammation serum cytokine levels (C-reactive protein > 0.2mg/dL). Atorvastatin (40mg/day) would be given to those who were allocated to the intervention group. The investigators will than follow up cardiac diastolic function by echocardiography and also the change of serum markers. The investigators would also genotype the inflammation-associated genes and their promoter region and find the association between genetic polymorphisms and the treatment effects of statins.

DETAILED DESCRIPTION:
We will evaluate left ventricular diastolic function noninvasively by echocardiography before and after the intervention. Exclusion criteria include coronary artery disease, significant valvular heart disease, cardiomyopathy, pericardial disease and renal insufficiency. We would like to enroll 50 cases and the same numbers of the controls. The inclusion criteria are subjects who underwent peritoneal dialysis at our hospital for more than 6 months with higher pro-inflammation serum cytokine levels (C-reactive protein > 0.2mg/dL). Atorvastatin (40mg/day) would be given to those who were allocated to the intervention group. We will than follow up cardiac diastolic function by echocardiography and also the change of serum markers. We would also genotype the inflammation-associated genes and their promoter region and find the association between genetic polymorphisms and the treatment effects of statins.

Patients population and Monitoring The study population will consist of patients with CAPD and DHF (NYHA Class II-IV), aged 18 years or older without reduced systolic function, defined as left ventricular EF ≤ 45%, Patients fulfilling the inclusion and exclusion criteria will be randomized in a 1:1 ratio into the study from the single medical centers.

Inclusion criteria:

1. Outpatients ≥ 20 year of age, male or female with essential hypertension
2. Patients must be on a stable condition of CAPD for at least 6 months.

Exclusion Criteria:

1. History of hypersensitivity to any of the study drugs.
2. Current acute decompensated HF (exacerbation of chronic HF manifested by signs & symptoms that may require IV therapy).
3. Acute coronary syndrome, stroke, transient ischemic attack, cardiac, carotid or major vascular surgery, percutaneous coronary intervention (PCI) or carotid angioplasty, within the past 3 months prior to visit 1.
4. Coronary or carotid artery disease likely to require surgical or percutaneous intervention within the 6 months after Visit 1.
5. Right heart failure due to severe pulmonary disease.
6. Diagnosis of peripartum or chemotherapy induced cardiomyopathy within the 12 months prior to visit 1.
7. Patients with a history of heart transplant or who are on a transplant list or with left ventricular assistance device (LVAD device).
8. Documented ventricular arrhythmia with syncopal episodes within past 3 months, prior to visit 1, that is untreated.
9. Symptomatic bradycardia or second or third degree heart block without a pacemaker.
10. Implantation of a CRT (cardiac resynchronization therapy) device within the prior 3 months from visit 1 or intent to implant a CRT device.
11. Presence of hemodynamically significant mitral and/or aortic valve disease, except mitral regurgitation secondary to left ventricular dilatation.
12. Presence of other hemodynamically significant obstructive lesions of left ventricular outflow tract, including aortic and sub-aortic stenosis.
13. Severe primary pulmonary, renal or hepatic disease judged by physicians.
14. Presence of any other disease with a life expectancy of < 1 year.
15. Chronic long-term requirement for NSAIDs (high dose) or COX2 inhibitors, with the exception of aspirin at doses used for CV prophylaxis (≤325 mg o.d.).
16. Subjects are now breast feeding, get pregnant or will be pregnant within 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients ≥ 20 year of age, male or female with essential hypertension
2. Patients must be on a stable condition of CAPD for at least 6 months.

Exclusion Criteria:

1. History of hypersensitivity to any of the study drugs.
2. Current acute decompensated HF (exacerbation of chronic HF manifested by signs & symptoms that may require IV therapy).
3. Acute coronary syndrome, stroke, transient ischemic attack, cardiac, carotid or major vascular surgery, percutaneous coronary intervention (PCI) or carotid angioplasty, within the past 3 months prior to visit 1.
4. Coronary or carotid artery disease likely to require surgical or percutaneous intervention within the 6 months after Visit 1.
5. Right heart failure due to severe pulmonary disease.
6. Diagnosis of peripartum or chemotherapy induced cardiomyopathy within the 12 months prior to visit 1.
7. Patients with a history of heart transplant or who are on a transplant list or with left ventricular assistance device (LVAD device).
8. Documented ventricular arrhythmia with syncopal episodes within past 3 months, prior to visit 1, that is untreated.
9. Symptomatic bradycardia or second or third degree heart block without a pacemaker.
10. Implantation of a CRT (cardiac resynchronization therapy) device within the prior 3 months from visit 1 or intent to implant a CRT device.
11. Presence of hemodynamically significant mitral and/or aortic valve disease, except mitral regurgitation secondary to left ventricular dilatation.
12. Presence of other hemodynamically significant obstructive lesions of left ventricular outflow tract, including aortic and sub-aortic stenosis.
13. Severe primary pulmonary, renal or hepatic disease judged by physicians.
14. Presence of any other disease with a life expectancy of < 1 year.
15. Chronic long-term requirement for NSAIDs (high dose) or COX2 inhibitors, with the exception of aspirin at doses used for CV prophylaxis (≤325 mg o.d.).
16. Subjects are now breast feeding, get pregnant or will be pregnant within 6 months.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2011-11; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Left ventricular diastolic function | 1 year
  We will arrange UCG follow up to delineate the change of LV diastolic function after intervention

SECONDARY OUTCOMES:
Mortality | 1 year
  Total Mortality differences
Major cardiovascular events | 1 year
  Check the MACE differences
Side effects | 1 year
  Follow up the number of rhabdomyolyis, hepatitis

CONTACTS AND LOCATIONS:
Overall Officials: Cho-Kai Wu, MD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Wu CK, Yeh CF, Chiang JY, Lin TT, Wu YF, Chiang CK, Kao TW, Hung KY, Huang JW. Effects of atorvastatin treatment on left ventricular diastolic function in peritoneal dialysis patients-The ALEVENT clinical trial. J Clin Lipidol. 2017 May-Jun;11(3):657-666. doi: 10.1016/j.jacl.2017.02.016. Epub 2017 Mar 18. PMID 28506387